CLINICAL TRIAL: NCT04195685
Title: Neurofeedback Impact on Chronic Headache, Sleep and Attention Disorders Experienced by Veterans With Mild Traumatic Brain Injury
Brief Title: Neurofeedback Impact on Veterans With mTBI
Acronym: NFBVETmTBI
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: VA Office of Research and Development (U.S. Federal Agency)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: NURC-002-19S; CX00164501A2 (Other Grant/Funding Number: CSR&D)
Record Dates: First submitted 2019-12-06; First posted 2019-12-12 (Actual); Results first posted 2025-10-30 (Actual); Last update posted 2025-10-30 (Actual); Status verified 2025-10

CONDITIONS: Concussion; mTBI; Post-Concussive Symptoms; Chronic Headache; Chronic Insomnia; Chronic Attention Disorder
Keywords: Neurofeedback; Infra-Low Frequency Neurofeedback; Veterans; Integrative Health Treatment; mTBI; Concussion; Post-concussive Symptoms; Chronic Headaches; Chronic Insomnia; Chronic Attention Disorder; Quality of Life; Emotional Responses; PTSD; Depression
MeSH Terms: conditions — Brain Concussion; Post-Concussion Syndrome; Headache Disorders; Sleep Initiation and Maintenance Disorders; Stress Disorders, Post-Traumatic; Depression | interventions — Neurofeedback

STUDY DESIGN:
Intervention Model Description: The proposed study is a randomized controlled clinical trial using Neurofeedback (NFB) as the study intervention. The control group members will continue with their usual care and will receive a 15-minute phone call from an Investigator on a weekly basis to briefly discuss one of eight possible health topics (sleep hygiene, basic nutritional concepts, beverage choices, positive thinking, thought reframing, fitness, daily calming activity, and enhancement of focus strategies) that the treatment group would receive as a normal part of their NFB session. At the end of the Control group activities, the participant will enter the delayed intervention group. Twenty, one-hour, NFB training sessions will be provided to each participant in the intervention group by a trained NFB specialist over an 8-10-week period (up to 5-sessions but usually 3 sessions a week).
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- NFB Intervention and Delayed Intervention (Experimental): The NFB system will read and interpret a participant's brain wave pattern which will be instantaneously fed back to the participant providing information, to which a participant can respond accordingly. The NFB specialist assumes a coaching role with people training on the NFB special use system to assist in the achievement of a focused relaxed state, which enhances the overall brain functioning. The significance and unique aspect of NFB is the direct impact on physiological dysregulation, which is the basis of this treatment approach. Twenty, one-hour, NFB training sessions will be provided to each participant in the intervention group and Delayed intervention group (those participants who completed the Control Group activities) by a trained NFB specialist over an 8-10-week period. Participants in the intervention group will receive up to 5-sessions but usually 3 sessions a week
  Interventions: Procedure: Neurofeedback (NFB)
- Control Group (No Intervention): Participants in the control group will continue with their usual treatment and will receive a 15-minute call once a week for eight weeks from an Investigator on a health topic. This will help to keep members of the control group engaged in the project and receive the same information that is offered to the intervention group members. The health topics that are generally discussed during NFB sessions include sleep hygiene, basic nutritional concepts, beverage choices, positive thinking, thought reframing, fitness, daily calming activity, and enhancement of focus strategies.

INTERVENTIONS:
Procedure: Neurofeedback (NFB) — Participants are seated in a comfortable chair and have common EEG electrodes with a pre-application of EEG adhesion conductive paste placed on scalp. The participant will receive coaching as they look at the game training screen and focus on the image. The game training screen provides almost instantaneous feedback (within 200 milliseconds) to participants about brain functioning. Twenty, one-hour, NFB training sessions will be provided by a trained NFB specialist over an 8-10-week period with up to 5-sessions but usually 3 sessions a week. The specific NFB special use system that will be used is the Cygnet NFB System from Bee Medic Corporation. The latest technological advances in this system has enabled training frequencies in the infra-low frequency range as well as in all other relevant frequency ranges which is a breakthrough capacity not available on any other NFB system. This will enable the individualized training to the person's brain training preference.
  Other Names: EEG Biofeedback, Neurotherapy
  Arms: NFB Intervention and Delayed Intervention

SUMMARY:
This study will evaluate neurofeedback (NFB) training as a low risk, non-invasive, effective treatment for Veterans diagnosed with mild traumatic brain injury (mTBI) and experiencing chronic post-concussive symptoms (PCSs). Participants will be randomized into the intervention or control group. Groups will be compared on primary measures of headache, insomnia and attention. Other outcomes of interest include post-traumatic stress symptoms, depression, quality of life and other measures of well-being.

DETAILED DESCRIPTION:
This study will evaluate neurofeedback (NFB) training as a low risk, non-invasive, effective treatment for Veterans diagnosed with mild traumatic brain injury (mTBI) and experiencing chronic post-concussive symptoms (PCSs). Participants will be randomized into the intervention or control group. Groups will be compared on primary measures of headache, insomnia and attention. Other outcomes of interest include post-traumatic stress symptoms, depression, quality of life and other measures of well-being.

Both the intervention and control group will participate in four assessment sessions. The assessment sessions will occur at the beginning of the study, at 4-6 weeks, at 8-10 weeks, and 2-months later. Participation in this research will last about 4 months. Those in the control group will be offered neurofeedback treatment, extending their participation time by 4 months (8 months total participation).

ELIGIBILITY:
Inclusion Criteria:

* Male and non-pregnant female OEF-OIF-OND Veterans diagnosed with mTBI ages 18 to 65
* Complaints of chronic headaches, insomnia, and attention difficulties
* Able to read and write English
* Able to comprehend what they read
* Able to follow directions

Exclusion Criteria:

* Pregnant female Veteran
* Non OEF-OIF-OND Veteran who is diagnosed with mTBI
* Under the age of 18 or over the age of 65
* Severe TBI
* Impaired decision-making capacity
* Unable to comply with study visit schedule
* Suicide Intent as indicated by a positive response to questions 3, 4, 5, or 8 on the Columbia Suicide Severity Rating Scale (C-SSRS) secondary screen

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 87 (Actual)
Dates: Start 2021-03-16 (Actual); Primary Completion 2024-09-16 (Actual); Study Completion 2025-02-10 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Judy M Carlson, EdD, Principal Investigator — VA Pacific Islands Health Care System, Honolulu, HI
Locations (1):
- VA Pacific Islands Health Care System, Honolulu, HI, Honolulu, Hawaii, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Moshkani Farahani D, Tavallaie SA, Ahmadi K, Fathi Ashtiani A. Comparison of neurofeedback and transcutaneous electrical nerve stimulation efficacy on treatment of primary headaches: a randomized controlled clinical trial. Iran Red Crescent Med J. 2014 Aug;16(8):e17799. doi: 10.5812/ircmj.17799. Epub 2014 Aug 5. PMID 25389484
- [Background] Sayer NA, Rettmann NA, Carlson KF, Bernardy N, Sigford BJ, Hamblen JL, Friedman MJ. Veterans with history of mild traumatic brain injury and posttraumatic stress disorder: challenges from provider perspective. J Rehabil Res Dev. 2009;46(6):703-16. doi: 10.1682/jrrd.2009.01.0008. PMID 20104400
- [Background] Morissette SB, Woodward M, Kimbrel NA, Meyer EC, Kruse MI, Dolan S, Gulliver SB. Deployment-related TBI, persistent postconcussive symptoms, PTSD, and depression in OEF/OIF veterans. Rehabil Psychol. 2011 Nov;56(4):340-50. doi: 10.1037/a0025462. PMID 22121940
- [Background] Lange RT, Brickell TA, Ivins B, Vanderploeg RD, French LM. Variable, not always persistent, postconcussion symptoms after mild TBI in U.S. military service members: a five-year cross-sectional outcome study. J Neurotrauma. 2013 Jun 1;30(11):958-69. doi: 10.1089/neu.2012.2743. Epub 2013 Jun 5. PMID 23205671
- [Background] Shandera-Ochsner AL, Berry DT, Harp JP, Edmundson M, Graue LO, Roach A, High WM Jr. Neuropsychological effects of self-reported deployment-related mild TBI and current PTSD in OIF/OEF veterans. Clin Neuropsychol. 2013;27(6):881-907. doi: 10.1080/13854046.2013.802017. Epub 2013 Jun 11. PMID 23755991

RESULTS

PARTICIPANT FLOW:
Groups:
- NFB Intervention: The NFB system will read and interpret a participant's brain wave pattern which will be instantaneously fed back to the participant providing information, to which a participant can respond accordingly. The NFB specialist assumes a coaching role with people training on the NFB special use system to assist in the achievement of a focused relaxed state, which enhances the overall brain functioning. The significance and unique aspect of NFB is the direct impact on physiological dysregulation, which is the basis of this treatment approach. Twenty, one-hour, NFB training sessions will be provided to each participant in the intervention group and Delayed intervention group (those participants who completed the Control Group activities) by a trained NFB specialist over an 8-10-week period. Participants in the intervention group will receive up to 5-sessions but usually 3 sessions a week
  Neurofeedback (NFB): Participants are seated in a comfortable chair and have common EEG electrodes with a pre-application of EEG adhesion conductive paste placed on scalp. The participant will receive coaching as they look at the game training screen and focus on the image. The game training screen provides almost instantaneous feedback (within 200 milliseconds) to participants about brain functioning. The Cygnet NFB System will be used, which enables training frequencies in the infra-low frequency range. This will enable the individualized training to the person's brain training preference.
Period: Overall Study
Arm/Group | NFB Intervention | Control Group
Started | 43 | 44
Mid-treatment (Mid-treatment assessment occurred after 10th session of neurofeedback or after 4th phone call in the control procedures.) | 39 | 39
Post-treatment (Post-treatment assessment occurred after 20th (last) session of neurofeedback or 8th (last) phone call in the control procedures.) | 37 | 38
2-month Follow up (2-month follow up assessment occurred approximately 2 months after the date of the post-treatment assessment.) | 36 | 38
Completed | 36 | 38
Not Completed | 7 | 6
Not completed — Withdrawal by Subject | 6 | 2
Not completed — Lost to Follow-up | 1 | 4

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | NFB Intervention | Control Group | Total
Number analyzed (Participants) | 43 | 44 | 87
Age, Continuous [Mean (Standard Deviation); unit: years] | 45.8 (7.7) | 45.0 (8.4) | 45.4 (8.1)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 6 | 8 | 14
  Male | 37 | 36 | 73
Race/Ethnicity, Customized [Count of Participants; unit: Participants]
  Self-identified ethnicity: African/Black | 4 | 8 | 12
  Self-identified ethnicity: European/Caucasian | 12 | 10 | 22
  Self-identified ethnicity: Asian | 4 | 5 | 9
  Self-identified ethnicity: Native American | 1 | 0 | 1
  Self-identified ethnicity: Hispanic | 9 | 3 | 12
  Self-identified ethnicity: Hawaiian/Pacific Islander | 3 | 1 | 4
  Self-identified ethnicity: More than one ethnicity | 10 | 15 | 25
  Self-identified ethnicity: Refused/Unknown | 0 | 2 | 2
Headache Impact Tool (HIT-6) [Mean (Standard Deviation); unit: score on a scale] — 6-item measure, score range 36-78. Higher score suggests greater impact
  score on a scale | 61.7 (8.8) | 62.8 (5.6) | 62.3 (7.2)
NEUROQOLTBI Headache Tool [Mean (Standard Deviation); unit: score on a scale] — 10-item form, scores range from: 10-50; Lower score suggests less headache pain
  score on a scale | 32.0 (10.9) | 31.7 (8.5) | 31.9 (9.7)
Insomnia Severity Index (ISI) [Mean (Standard Deviation); unit: score on a scale] — 7-item form, score range: 0-28. Higher scores suggest greater severity
  score on a scale | 19.4 (4.6) | 18.5 (5.6) | 19.0 (5.1)
NEUROQOLTBI Sleep Disturbance [Mean (Standard Deviation); unit: score on a scale] — 8-item form, score range: 8-40. Higher score suggest greater impact
  score on a scale | 25.8 (6.7) | 26.0 (6.0) | 25.9 (6.4)
QIK test accuracy index [Mean (Standard Deviation); unit: score on a scale] | 232.9 (39.0) | 241.3 (44.9) | 237.1 (42.0)
Quality of Life after Brain Injury (QOLIBRI) [Mean (Standard Deviation); unit: score on a scale] — 37-item form, score range: 0-100. Higher score suggests higher quality of life
  score on a scale | 46.3 (17.3) | 46.3 (17.2) | 46.3 (17.3)
NEUROQOLTBI Satisfaction with roles and activities [Mean (Standard Deviation); unit: score on a scale] — 8-item form, score range: 8-40. Higher score suggests more satisfaction.
  score on a scale | 23.1 (7.4) | 21.9 (6.1) | 22.5 (6.8)
NEUROQOLTBI Ability to participate in social roles and activities [Mean (Standard Deviation); unit: score on a scale] — 8-item form, score range 8-40. Higher score suggest better participation ability
  score on a scale | 25.0 (6.8) | 24.4 (5.7) | 24.7 (6.3)
General Symptom Scale (GSI) [Mean (Standard Deviation); unit: score on a scale] — 116-item form, score range 0-464. Higher score suggests more severity or increased frequency
  score on a scale | 166.6 (83.7) | 156.7 (54.0) | 161.7 (68.9)
Depression, Anxiety and Stress Scale (DASS21) [Mean (Standard Deviation); unit: score on a scale] — 21 item form, score range: 0-63. Higher score suggests more distress.
  score on a scale | 24.2 (15.3) | 23.9 (12.4) | 24.1 (13.9)
Post-Traumatic Stress Disorder Checklist (PCL-5) [Mean (Standard Deviation); unit: score on a scale] — 20-item form, score range 0-80. Higher score suggests greater stress
  score on a scale | 40.7 (20.4) | 40.9 (18.7) | 40.8 (19.6)
Patient Health Questionnaire-Depression (PHQ9) [Mean (Standard Deviation); unit: score on a scale] — 9-item form, score range: 0-27. Higher score suggests greater impact
  score on a scale | 14.3 (6.6) | 14.3 (5.7) | 14.3 (6.2)
NEUROQOLTBI Positive affect and wellbeing [Mean (Standard Deviation); unit: score on a scale] — 9-item form, score range: 9-45. Higher score suggests better health
  score on a scale | 29.9 (8.2) | 29.8 (5.8) | 29.9 (7.0)

OUTCOME MEASURES:

1. Primary Outcome: Headache Impact Test (HIT-6)
Description: The HIT-6 is a 6-question tool designed to describe and communicate the way people feel and what they cannot do because of their headache. (6 questions, 3 min) Scores vary from 36 - 78. Higher score worse outcome.
Time Frame: Change from baseline midtreatment at 4-6 weeks, change from baseline endpoint at 8-10 weeks, and change from baseline at 2 month follow-up
Population: Primary analyses were intention to treat, which included all participants assigned to either group. Missing data were addressed using a multiple imputation approach.
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | NFB Intervention | Control Group
Number analyzed (Participants) | 43 | 44
score on a scale
  Mid-treatment | 53.2 (9.8) | 61.4 (6.6)
  Post-treatment | 49.2 (10.4) | 60.9 (7.4)
  2-month follow-up | 52.2 (11.5) | 62.6 (8.7)
Statistical Analysis 1: Comparison: NFB Intervention vs Control Group; The primary endpoint was evaluated by assessing the change in severity scores from baseline to the end of treatment, comparing the NFB and control groups. A two-sample t-test was used to test the mean change in severity scores between treatment arms. Statistical tests were two-sided with a 5% significance level (Type I error rate); Test type: Other; p < .0001, t-test, 2 sided; Mean Difference (Final Values) = 10.7, 95% CI 2-sided [7.0 to 14.4]

2. Primary Outcome: NEUROQOLTBI Headache Pain Short Form
Description: Developed as part of NIH Toolbox NEUROQOL TBI. It is comprised of 10 questions related to the nature and response to headaches. (10 items, 5 minutes). Score range 10-50. Higher scores suggest worse outcome.
Time Frame: as for outcome 1
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | NFB Intervention | Control Group
Number analyzed (Participants) | 43 | 44
score on a scale
  Mid-treatment | 21.3 (11.3) | 28.5 (10.2)
  Post-treatment | 18.9 (11.2) | 28.0 (11.6)
  2-month follow-up | 23.1 (13.0) | 32.4 (11.3)
Statistical Analysis 1: Comparison: NFB Intervention vs Control Group; [analysis description as in outcome 1, analysis 1]; Test type: Other; p < .0001, t-test, 2 sided; Mean Difference (Final Values) = 9.5, 95% CI 2-sided [4.9 to 14.0]

3. Primary Outcome: Insomnia Severity Index (ISI)
Description: Seven question self-report instrument used to quantify perceived current insomnia. Targets past week's symptoms and daytime consequences consistent with DSM-IV criteria. (7 items, 5 min) Scores vary from 0 - 28. Higher score worse outcome.
Time Frame: as for outcome 1
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | NFB Intervention | Control Group
Number analyzed (Participants) | 43 | 44
score on a scale
  Mid-treatment | 11.5 (7.1) | 17.2 (6.2)
  Post-treatment | 7.7 (7.3) | 17.1 (6.3)
  2-month follow-up | 10.2 (7.9) | 17.0 (7.0)
Statistical Analysis 1: Comparison: NFB Intervention vs Control Group; [analysis description as in outcome 1, analysis 1]; Test type: Other; p < .0001, t-test, 2 sided; Mean Difference (Final Values) = 10.3, 95% CI 2-sided [7.4 to 13.2]

4. Primary Outcome: NEUROQOLTBI Sleep Disturbance Short Form
Description: Developed as part of NIH Toolbox NEUROQOL TBI. It is comprised of 8 questions related to the sleep experience and impact. (8 items, 5 minutes). Score range: 8-40. Higher scores suggest worse outcome.
Time Frame: as for outcome 1
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | NFB Intervention | Control Group
Number analyzed (Participants) | 43 | 44
score on a scale
  Mid-treatment | 29.2 (8.1) | 22.0 (7.3)
  Post-treatment | 31.2 (9.9) | 22.3 (8.0)
  2-month follow-up | 28.6 (9.9) | 22.7 (7.8)
Statistical Analysis 1: Comparison: NFB Intervention vs Control Group; [analysis description as in outcome 1, analysis 1]; Test type: Other; p < .0001, t-test, 2 sided; Mean Difference (Final Values) = 7.4, 95% CI 2-sided [4.2 to 10.6]

5. Primary Outcome: QIKtest Continuous Performance Test - Accuracy Index
Description: Computerized visual performance test to assess attention and impulse control, speed and consistency of response. Specifically intended for use by neurofeedback clinicians. (21 min). Higher scores indicate better performance. Score range: 165-420.
Time Frame: as for outcome 1
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | NFB Intervention | Control Group
Number analyzed (Participants) | 43 | 44
score on a scale
  Mid-treatment | 252.0 (41.9) | 241.6 (50.1)
  Post-treatment | 271.4 (60.8) | 247.3 (58.7)
  2-month follow-up | 254.4 (48.4) | 256.8 (56.8)
Statistical Analysis 1: Comparison: NFB Intervention vs Control Group; [analysis description as in outcome 1, analysis 1]; Test type: Other; p = 0.0022, t-test, 2 sided; Mean Difference (Final Values) = -32.5, 95% CI 2-sided [-53.3 to -11.7]

6. Primary Outcome: Quality of Life After Brain Injury (QOLIBRI)
Description: A 37-item instrument consisting of 6 scales measuring cognition, self, daily life and autonomy, social relationships, emotions, and physical problems. Designed to measure quality of life specific for TBI. (37 items, 15 min). Score range: 0-100. Higher score suggests better outcome.
Time Frame: as for outcome 1
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | NFB Intervention | Control Group
Number analyzed (Participants) | 43 | 44
score on a scale
  Mid-treatment | 127.4 (32.6) | 106.8 (27.4)
  Post-treatment | 139.8 (36.3) | 107.6 (31.0)
  2-month follow-up | 133.8 (38.8) | 108.6 (30.3)
Statistical Analysis 1: Comparison: NFB Intervention vs Control Group; [analysis description as in outcome 1, analysis 1]; Test type: Other; p < .0001, t-test, 2 sided; Mean Difference (Final Values) = -32.2, 95% CI 2-sided [-45.0 to -19.4]

7. Primary Outcome: NEUROQOLTBI Satisfaction With Social Roles and Activities Short Form
Description: Developed as part of NIH Toolbox NEUROQOL TBI. It is comprised of 10 questions related to level of satisfaction with life roles and activities. (10 items, 5 min). Score range: 8-40. Higher score suggests better outcome.
Time Frame: as for outcome 1
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | NFB Intervention | Control Group
Number analyzed (Participants) | 43 | 44
score on a scale
  Mid-treatment | 33.5 (7.6) | 30.0 (6.8)
  Post-treatment | 35.4 (8.7) | 31.2 (7.6)
  2-month follow-up | 34.8 (8.5) | 30.0 (7.5)
Statistical Analysis 1: Comparison: NFB Intervention vs Control Group; [analysis description as in outcome 1, analysis 1]; Test type: Other; p = 0.0002, t-test, 2 sided; Mean Difference (Final Values) = -7.3, 95% CI 2-sided [-11.1 to -3.4]

8. Primary Outcome: NEUROQOLTBI Ability to Participate in Social Roles and Activities Short Form
Description: Developed as part of NIH Toolbox NEUROQOL TBI. It is comprised of 10 questions related to level of ability to do life roles and activities. (10 items, 5 min). Score range 8-40. Higher score suggests better outcome.
Time Frame: as for outcome 1
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | NFB Intervention | Control Group
Number analyzed (Participants) | 43 | 44
score on a scale
  Mid-treatment | 29.1 (7.3) | 24.7 (5.8)
  Post-treatment | 31.0 (8.2) | 24.2 (6.7)
  2-month follow-up | 29.7 (8.4) | 24.8 (6.6)
Statistical Analysis 1: Comparison: NFB Intervention vs Control Group; [analysis description as in outcome 1, analysis 1]; Test type: Other; p < .0001, t-test, 2 sided; Mean Difference (Final Values) = -6.2, 95% CI 2-sided [-9.0 to -3.4]

9. Primary Outcome: NEUROQOLTBI Positive Affect and Well-being-short Form
Description: Developed as part of NIH Toolbox NEUROQOL TBI. It is comprised of 10 questions related to level of positive attitude and sense of well-being (9 items, 5 min). Score range: 9-45. Higher score better outcome.
Time Frame: as for outcome 1
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | NFB Intervention | Control Group
Number analyzed (Participants) | 43 | 44
score on a scale
  Mid-treatment | 33.5 (7.3) | 30.2 (6.8)
  Post-treatment | 35.5 (8.2) | 31.0 (7.0)
  2-month follow-up | 34.7 (8.5) | 30.1 (7.1)
Statistical Analysis 1: Comparison: NFB Intervention vs Control Group; Test type: Other; p = 0.0033, t-test, 2 sided; Mean Difference (Final Values) = -4.5, 95% CI 2-sided [-7.4 to -1.5]

10. Secondary Outcome: Depression, Anxiety and Stress Scale 21 (DASS21)
Description: DASS21 is a set of three self-report scales designed to measure the negative emotional states of depression, anxiety and stress. Can be used as a single assessment of psychological distress (21 items, 10 min). Score varies from 0 - 63. Higher score suggests worse outcome.
Time Frame: as for outcome 1
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | NFB Intervention | Control Group
Number analyzed (Participants) | 43 | 44
score on a scale
  Mid-treatment | 12.0 (11.6) | 20.3 (12.4)
  Post-treatment | 10.2 (12.7) | 19.9 (13.4)
  2-month follow-up | 13.3 (13.9) | 23.1 (13.6)
Statistical Analysis 1: Comparison: NFB Intervention vs Control Group; [analysis description as in outcome 1, analysis 1]; Test type: Other; p = 0.0005, t-test, 2 sided; Mean Difference (Final Values) = 10.0, 95% CI 2-sided [4.4 to 15.6]

11. Secondary Outcome: Patient Health Questionnaire-9 (PHQ-9)
Description: PHQ-9 is a nine-item depression self-report module from the full Patient Health Questionnaire. Scores range from 0-27. (9 items, 2-5 min) Score varies from 0-27. Higher score suggests worse outcome.
Time Frame: as for outcome 1
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | NFB Intervention | Control Group
Number analyzed (Participants) | 43 | 44
score on a scale
  Mid-treatment | 8.2 (6.8) | 12.2 (6.2)
  Post-treatment | 5.7 (7.2) | 12.0 (6.7)
  2-month follow-up | 7.4 (7.5) | 13.1 (7.0)
Statistical Analysis 1: Comparison: NFB Intervention vs Control Group; [analysis description as in outcome 1, analysis 1]; Test type: Other; p < .0001, t-test, 2 sided; Mean Difference (Final Values) = 6.4, 95% CI 2-sided [3.5 to 9.2]

12. Secondary Outcome: Posttraumatic Stress Disorder Checklist (PCL-5)
Description: The PCL-5 is a 20-item questionnaire, corresponding to the DSM-5 symptom criteria for PTSD. The wording of PCL-5 items reflects both changes to existing symptoms and the addition of new symptoms in DSM-5. (20 items, 5-10 min) Score varies from 0-80. Higher score suggests worse outcome.
Time Frame: as for outcome 1
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | NFB Intervention | Control Group
Number analyzed (Participants) | 43 | 44
score on a scale
  Mid-treatment | 25.4 (19.3) | 35.7 (17.5)
  Post-treatment | 19.3 (20.2) | 33.7 (19.1)
  2-follow follow-up | 23.0 (21.0) | 37.1 (20.3)
Statistical Analysis 1: Comparison: NFB Intervention vs Control Group; [analysis description as in outcome 1, analysis 1]; Test type: Other; p = 0.0001, t-test, 2 sided; Mean Difference (Final Values) = 14.2, 95% CI 2-sided [7.1 to 21.4]

13. Secondary Outcome: General Symptom Inventory (GSI)
Description: Self-report instrument of symptoms in 7 categories including sleep, attention and learning, sensory, behavioral, emotional, physical, and pain (less than 10 min). Score varies from 0-464. Higher score suggests worse outcome.
Time Frame: as for outcome 1
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | NFB Intervention | Control Group
Number analyzed (Participants) | 43 | 44
score on a scale
  Mid-treatment | 108.7 (75.9) | 151.7 (61.0)
  Post-treatment | 81.3 (90.2) | 139.4 (73.4)
  2-month follow-up | 103.1 (97.9) | 150.4 (72.9)
Statistical Analysis 1: Comparison: NFB Intervention vs Control Group; [analysis description as in outcome 1, analysis 1]; Test type: Other; p < .0001, t-test, 2 sided; Mean Difference (Final Values) = 68.0, 95% CI 2-sided [36.9 to 99.2]

ADVERSE EVENTS:
Time Frame: Adverse event data were collected while the participant was actively involved in study procedures. Depending on randomized group membership, this was either baseline to 4 months (neurofeedback) or 8 months (control, later delayed intervention) for those who completed study procedures. Participants who withdrew were followed for adverse event data until their withdrawal date.
Groups:
- NFB Intervention: The NFB system will read and interpret a participant's brain wave pattern which will be instantaneously fed back to the participant providing information, to which a participant can respond accordingly. The NFB specialist assumes a coaching role with people training on the NFB special use system to assist in the achievement of a focused relaxed state, which enhances the overall brain functioning. The significance and unique aspect of NFB is the direct impact on physiological dysregulation, which is the basis of this treatment approach. Twenty, one-hour, NFB training sessions will be provided to each participant in the intervention group and Delayed intervention group (those participants who completed the Control Group activities) by a trained NFB specialist over an 8-10-week period. Participants in the intervention group will receive up to 5-sessions but usually 3 sessions a week
  Neurofeedback (NFB): Participants are seated in a comfortable chair and have common EEG electrodes with a pre-application of EEG adhesion conductive paste placed on scalp. The participant will receive coaching as they look at the game training screen and focus on the image. The game training screen provides almost instantaneous feedback (within 200 milliseconds) to participants about brain functioning. The Cygnet NFB System, which enables training frequencies in the infra-low frequency range will be used. This will enable the individualized training to the person's brain training preference.
- Control Group: Participants in the control group will continue with their usual treatment and will receive a 15-minute call once a week for eight weeks from an Investigator on a health topic. This will help to keep members of the control group engaged in the project and receive the same information that is offered to the intervention group members. The health topics that are generally discussed during NFB sessions include sleep hygiene, basic nutritional concepts, beverage choices, positive thinking, thought reframing, fitness, daily calming activity, and enhancement of focus strategies. Upon completion control group activities, participants had the option to receive the neurofeedback intervention. They then followed the NFB intervention protocol.
Arm/Group | NFB Intervention | Control Group
All-Cause Mortality (participants affected / at risk) | 0/43 | 0/44
Serious Adverse Events (participants affected / at risk) | 1/43 | 1/44
Other Adverse Events (participants affected / at risk) | 3/43 | 12/44
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | NFB Intervention (N=43) | Control Group (N=44)
Inpatient Hospitalization (Psychiatric disorders) | 1 (1) | 1 (1)
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | NFB Intervention (N=43) | Control Group (N=44)
Psychological (Psychiatric disorders) | 2 (2) | 1 (1) — description of new or exacerbating psychological symptoms
Medical (Infections and infestations) | 1 (1) | 2 (2) — any report of infection regardless of location
Medical (Surgical and medical procedures) | 0 (0) | 1 (1) — any outpatient surgical or medical procedure
Medical (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 6 (6) — includes COVID-19 diagnoses
Medical (Nervous system disorders) | 0 (0) | 1 (1)
Medical (Cardiac disorders) | 0 (0) | 1 (1)
Medical (General disorders) | 0 (0) | 1 (3) — includes AEs that cross multiple systems
Medical (Vascular disorders) | 0 (0) | 1 (1)
Medical (Eye disorders) | 0 (0) | 1 (1)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (2):
  • Study Protocol and Statistical Analysis Plan (2025-04-03): https://cdn.clinicaltrials.gov/large-docs/85/NCT04195685/Prot_SAP_001.pdf
  • Informed Consent Form (2023-06-13): https://cdn.clinicaltrials.gov/large-docs/85/NCT04195685/ICF_000.pdf